CLINICAL TRIAL: NCT06778811
Title: Clinical Study of Perioperative Sleep Disorders in Cardiac Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20240924-05
Record Dates: First submitted 2024-12-23; First posted 2025-01-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Sleep Wake Disorders; Esketamine and the Quality of Recovery; Dexmedetomidine
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dexmedetomidine group (Experimental): Intraoperative infusion of 0.3ug/kg/h dexmedetomidine
  Interventions: Drug: Intraoperative infusion of dexmedetomidine
- esketamine group (Experimental): Intraoperative infusion of 0.3mg/kg/h esketamine
  Interventions: Drug: Intraoperative infusion of esketamine
- control group (Placebo Comparator): Intraoperative infusion of equal volumes of saline
  Interventions: Drug: Saline control

INTERVENTIONS:
Drug: Intraoperative infusion of dexmedetomidine — Intraoperative infusion of 0.3ug/kg/h dexmedetomidine
  Arms: dexmedetomidine group
Drug: Intraoperative infusion of esketamine — Intraoperative infusion of 0.3mg/kg/h esketamine
  Arms: esketamine group
Drug: Saline control — Intraoperative infusion of equal volumes of saline
  Arms: control group

SUMMARY:
The aim of this clinical trial is to understand the effects of dexmedetomidine and esketamine on postoperative sleep in patients undergoing cardiac surgery. The main questions it aims to answer are:

Does dexmedetomidine or esketamine prevent the development of postoperative sleep disturbances? Which one works better? The researchers compared dexmedetomidine and esketamine with saline (a drug-free solvent) to see if dexmedetomidine and esketamine prevented the development of postoperative sleep disturbances.

Participants will:

1. Intraoperative continuous infusion of dexmedetomidine, esketamine or saline until the end of surgery
2. Postoperative sleep was assessed on the first and third postoperative days using a sleep rating scale

ELIGIBILITY:
Inclusion Criteria:

1. ASA class II-III, NYHA class I-III, EF ≥ 50%
2. Intended to perform cardiac surgery under extracorporeal circulation

Exclusion Criteria:

1. Patients undergoing second heart surgery
2. Patients with mental retardation, deafness, or other conditions that interfere with normal communication
3. Previous neurological or psychiatric disorders
4. Patients with a history of sleep disorders
5. Alcoholics, drug addicts, or psychotropic substance abusers
6. Significant hepatic or renal dysfunction affecting drug metabolism
7. Contraindication to the use of dexmedetomidine or esketamine.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 1, 3, 7days after surgery
  Assessment of sleep quality by the Athens Insomnia Scale (AIS) and smart wearable device

SECONDARY OUTCOMES:
postoperative pain | 24 hours and 48 hours after surgery
  Assessment of postoperative pain levels by Visual Analogue Scale（VAS），from 0 to 10, Higher scores mean more severe pain，VAS>4 means positive.
Record postoperative analgesic medications used and the amount used for postoperative pain | 24 hours and 48 hours after surgery
  Record postoperative analgesic medications used and the amount used
anxiety and depression assessment | 1,3 days after surgery
  Assessment of anxiety and depression levels by Hospital anxiety and depression scale (HADS)，0-7 is negative; 8-10 is mild; 11-14 is moderate; 15-21 is severe.
Postoperative complications | 48 hours after surgery
  including nausea and vomiting, dizziness, itching, nightmares and so on.
Postoperative delirium | from 1 day to 7 days after surgery
  Assessment of Postoperative delirium by Confusion Assessment Method (CAM)，scores > 21 is positive.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing First Hospital，Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No